CLINICAL TRIAL: NCT00676559
Title: Combined aPproach to Treatment Using Ranibizumab and Efalizumab for Diabetic Macular Edema Study: The CAPTURE DME Study
Acronym: CAPTURE
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Unrelated serious adverse events involving one of the proposed medications
Sponsor: Johns Hopkins University (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Genentech, Inc. (Industry)
Responsible Party: Quan Dong Nguyen, MD, MSc, Johns Hopkins University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NA 00015499
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic; Macular; Edema; DME; Clinically Significant Macular Edema (CSME)
MeSH Terms: conditions — Edema | interventions — efalizumab; Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): Efalizumab 1 mg/kg weekly subcutaneous self-administered injections for 48 weeks.
  Interventions: Drug: Efalizumab
- Group 2 (Experimental): Ranibizumab 0.5 mg intravitreal injections monthly for three months followed by criteria-guided monthly injections through Month 11 (inclusive).
  Interventions: Drug: Ranibizumab
- Group 3 (Experimental): Efalizumab 1 mg/kg weekly subcutaneous self-administered injections for 48 weeks in combination with ranibizumab 0.5 mg intravitreal injections monthly for three months followed by criteria-guided monthly injections through Month 11 (inclusive).
  Interventions: Drug: Efalizumab; Drug: Ranibizumab

INTERVENTIONS:
Drug: Efalizumab — Efalizumab 1 mg/kg weekly subcutaneous self-administered injections for 48 weeks.
  Other Names: Raptiva
  Arms: Group 1; Group 3
Drug: Ranibizumab — Ranibizumab 0.5 mg intravitreal injections monthly for three months followed by criteria-guided monthly injections through Month 11 (inclusive).
  Other Names: Lucentis
  Arms: Group 2; Group 3

SUMMARY:
This study looks to continue the study of anti-vegf therapy in patients with macular edema, and compare it to an anti-inflammatory therapy and a combined Anti-vegf and anti-inflammatory.

DETAILED DESCRIPTION:
Cell adhesion molecules are key mediators of inflammatory processes, which have been shown to play a role in the pathogenesis of diabetic retinopathy . Efalizumab inhibits the binding of leukocyte function-associated antigen-1 (LFA-1) to intercellular adhesion molecule-1 (ICAM-1) thereby inhibiting the adhesion of leukocytes to other cell types.

Clinical studies have demonstrated the bioactivities of intravitreal ranibizumab, a Vascular endothelial growth factor (VEGF) antagonist, in reducing retinal thickness and improving visual acuity in patients with diabetic macular edema (DME).

The objective of the CAPTURE Study is to assess the safety and tolerability of efalizumab, administered subcutaneously as a weekly (1 mg/kg) dose, compared to and in combination with ranibizumab, administered intravitreally (0.5 mg), in the treatment of DME.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent and authorization of use and disclosure of protected health information
* 18 years of Age
* Diagnosis of diabetes mellitus (type 1 or type 2)
* Serum HbA1c 5.5% within 12 months of randomization
* Retinal thickening (diabetic macular edema) involving the center of the fovea
* Diagnosis must be confirmed by fluorescein angiography and OCT images over 250
* Best corrected visual acuity score in the study eye of 20/40 to 20/320
* If a female of childbearing potential, a negative pregnancy test and commitment to the use of at least two forms of effective contraception.
* If a non-sterile male, commitment to the use of two forms of effective contraception.
* Demonstrate understanding of and ability to perform weekly self sub-cutaneous injections.

Exclusion Criteria:

* Panretinal or macular photocoagulation within 3 months of study entry in the study eye
* Use of intraocular or periocular injection of steroids in the study eye within 3 months of study entry
* Previous participation in a study and receipt of anti-angiogenic drugs (pegaptanib sodium, ranibizumab, bevacizumab, anecortave acetate, protein kinase C inhibitor, etc.) within 2 months of study entry
* Current or history of prior treatment of psoriasis with subcutaneous efalizumab within 6 months of study entry

  * Proliferative diabetic retinopathy in the study eye, with the exceptions of
  * inactive, fibrotic proliferative diabetic retinopathy that has regressed following pan-retinal laser photocoagulation OR
  * tufts of neovascularization elsewhere (NVE) less than one disc area with no vitreous hemorrhage
  * Vitreomacular traction or epiretinal membrane in the study eye
  * Structural damage to the center of the macula in the study eye likely to preclude improvement in visual acuity following the resolution of macular edema.
  * Concurrent disease in the study eye that could compromise visual acuity or require medical or surgical intervention during the first 6-months.
  * Cataract surgery in the study eye within 3 months of study entry; (YAG) laser capsulotomy within 1 month of study entry; or any other intraocular surgery within 3 months preceding Day 0.
  * History of vitreoretinal surgery in the study eye within 3 months of study entry
  * Uncontrolled glaucoma .
  * Blood pressure exceeding 180/100 (sitting) during the screening period
  * Uncontrolled diabetes mellitus, as evidenced by glycosylated hemoglobin > or = 13%(HbA1c) value
  * Renal failure requiring dialysis or renal transplant
  * Premenopausal women unwilling to commit to adequate contraception
  * History of other diseases or finding giving reasonable suspicion of a disease or condition that contraindicates the use an investigational drug, might affect interpretation of the results of the study, or render the subject at high risk from treatment complications
  * International Normalized Ratio (INR) > or = 3.0 (e.g. due to current treatment with warfarin).
  * History of cerebral vascular accident, myocardial infarction, transient ischemic attacks within 6 months of study enrollment.
  * Have a history of hypersensitivity to efalizumab
  * Have a history of ongoing uncontrolled serious bacterial, viral, fungal, or atypical mycobacterial infection. Have a history of opportunistic infections.
  * Have the presence or history of malignancy, including lymphoproliferative disorders.
  * Have a history of thrombocytopenia, clinically significant hemolytic anemia, or unexplained anemia
  * Have a platelet count < 100,000 cells/microliter (uL)
  * Inability to comply
  * Patients receiving immunosuppressive agents
  * All acellular, live and live-attenuated vaccines are excluded from 14 days prior to the first dose of efalizumab until a minimum of 4 weeks after the last dose of efalizumab
  * Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated.
  * Participation in another simultaneous medical investigation or trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2009-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of efalizumab, compared to and in combination with ranibizumab, measuring the frequency and severity of adverse events. | 6 mos

SECONDARY OUTCOMES:
To measure the mean change from Baseline to Month 6 and Month 12 in Best correct visual acuity (BCVA) | 6 and 12 mos.
To evaluate the anatomic retinal changes as assessed by color fundus photography, fluorescein angiography, and Optical Coherence Tomography (OCT) | 6 mos and 12 mos

CONTACTS AND LOCATIONS:
Overall Officials: Quan Dong Nguyen, MD, MSc, Study Director — Johns Hopkins University; Diana V Do, MD, Principal Investigator — Johns Hopkins University
Locations (10):
- United States (10):
  - Diego H. Calonje, M.D., P.C., Tucson, Arizona
  - Sharp Rees-Stealy Medical Group, San Diego, California
  - Retina Macula Institute, Torrance, California
  - Retina Associates of Maine, Bangor, Maine
  - Retina Center of Maine, South Portland, Maine
  - Wilmer Eye Institute at the Johns Hopkins University, Baltimore, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Eye Care Specialists, Kingston, Pennsylvania
  - Texas Retina Associates, Arlington, Texas
  - University of Utah, Salt Lake City, Utah